CLINICAL TRIAL: NCT00569673
Title: A Phase II Evaluation of Docetaxel (NSC #628503) Plus Trabectedin (Yondelis®), R279741, IND # 101018) With Growth Factor Support in the Third-Line Treatment of Recurrent or Persistent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Docetaxel, Trabectedin, and G-CSF or Pegfilgrastim in Treating Patients With Recurrent or Persistent Ovarian Epithelial Cancer, Primary Peritoneal Cavity Cancer, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Masking: None | Purpose: Treatment
Other Study IDs: GOG-0186F; GOG-0186F; CDR0000577866
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2014-05

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; fallopian tube cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Filgrastim; pegfilgrastim; Docetaxel; Trabectedin

INTERVENTIONS:
Biological: filgrastim
Biological: pegfilgrastim
Drug: docetaxel
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel and trabectedin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Colony-stimulating factors, such as G-CSF and pegfilgrastim, may help the immune system recover from the side effects of chemotherapy. Giving combination chemotherapy together with G-CSF or pegfilgrastim may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects and how well giving docetaxel and trabectedin together with G-CSF or pegfilgrastim works in treating patients with recurrent or persistent ovarian epithelial cancer, fallopian tube cancer, or primary peritoneal cavity cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the antitumor activity of docetaxel plus trabectedin in patients with persistent or recurrent ovarian epithelial, fallopian tube, or primary peritoneal cavity cancer primarily through the frequency of objective tumor responses.
* To determine the nature and degree of toxicity of docetaxel plus trabectedin in this cohort of patients.

Secondary

* To estimate the progression-free survival and overall survival of patients treated with docetaxel and trabectedin.

OUTLINE: Patients receive docetaxel IV over 1 hour and trabectedin IV over 3 hours on day 1. Patients also receive pegfilgrastim subcutaneously (SC) on day 1 OR filgrastim (G-CSF) IV over 15-30 minutes or SC once daily beginning on day 1 and continuing until blood counts recover. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed ovarian epithelial, fallopian tube, or primary peritoneal cavity carcinoma

  * Recurrent or persistent disease
* Measurable disease, defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest dimension to be recorded) ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have at least 1 "target lesion" to be used to assess response on this protocol as defined by RECIST criteria

  * Tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Must have had 1 prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound and the initial treatment may have included high-dose therapy, consolidation, or extended therapy administered after surgical or non-surgical assessment

  * Patients are allowed, but not required to receive, 2 additional cytotoxic regimens for management of recurrent or persistent disease with no more than 1 non-platinum, non-taxane regimen
  * Patients who have received only 1 prior cytotoxic regimen (platinum-based regimen for management of primary disease), must meet 1 of the following criteria:

    * Platinum-free interval of < 12 months
    * Progressed during platinum-based therapy
    * Persistent disease after a platinum-based therapy
* Not eligible for a higher priority GOG protocol (i.e., any active GOG Phase III protocol for the same patient population)

PATIENT CHARACTERISTICS:

* GOG performance status (PS) 0-2 or after receiving 1 prior treatment regimen (GOG PS 0-1 after receiving 2 or more prior regimens)
* Platelet count ≥ 100,000/mm³
* ANC count ≥ 1,500/mm³
* Hemoglobin > 9 g/dL
* Creatinine ≤ 1.5 times upper limit normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* CPK normal
* Bilirubin or direct bilirubin normal
* Alkaline phosphatase normal
* Neuropathy (sensory and motor) ≤ grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics (except for uncomplicated UTI)
* No other invasive malignancy within the past 5 years, except nonmelanoma skin cancer
* No known active liver disease or hepatitis
* Willing and able to have a central venous catheter

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from effects of recent surgery, radiotherapy, or chemotherapy
* At least 1 week since prior hormonal therapy directed at the malignant tumor

  * Continuation of hormone replacement therapy allowed
* At least 3 weeks since other prior therapy, including biological and immunological therapy directed at the tumor
* Chimeric or human or humanized monoclonal antibodies must be discontinued for at least 6 weeks prior to study entry
* No investigational therapy within the past 30 days
* No prior therapy with docetaxel and/or trabectedin
* No radiation to more than 25% of marrow-bearing areas
* No prior cancer treatment that contraindicates protocol therapy

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-03; Primary Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley J. Monk, MD, Study Chair — Chao Family Comprehensive Cancer Center; Kristine M. Zanotti, MD — MacDonald Physicians, Incorporated at University MacDonald Womens Hospital
Locations (37):
- United States (37):
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Carilion Gynecologic Oncology Associates, Roanoke, Virginia
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

REFERENCES:
- [Result] Monk BJ, Sill MW, Hanjani P, Edwards R, Rotmensch J, De Geest K, Bonebrake AJ, Walker JL. Docetaxel plus trabectedin appears active in recurrent or persistent ovarian and primary peritoneal cancer after up to three prior regimens: a phase II study of the Gynecologic Oncology Group. Gynecol Oncol. 2011 Mar;120(3):459-63. doi: 10.1016/j.ygyno.2010.11.012. Epub 2010 Dec 7. PMID 21144560
- [Result] Monk, M BJ, Sill M, Walker JL, et al.: Activity of docetaxel plus trabectedin in recurrent or persistent ovarian and primary peritoneal cancer: A phase II study of the Gynecologic Oncology Group (GOG). [Abstract] J Clin Oncol 28 (Suppl 15): A-5046, 2010.

RESULTS

PARTICIPANT FLOW:
Groups:
- Docetaxel Plus Trabectedin: Docetaxel 60 mg/m2 IV over 1 hour followed by trabectedin (YONDELIS"µ, R279741) formerly referred to as, ET-743) 1.1 mg/m2 over 3 hours with Filgrastim (G-CSF, NSC #614629), Pegfilgrastim (G-CSF, NSC #725961) or Sargramostim (GM-CSF, NSC #613795) every 3 weeks (one cycle) until disease progression or adverse effects prohibit further therapy.
Period: Overall Study
Arm/Group | Docetaxel Plus Trabectedin
Started | 71 (Total number participants enrolled on study)
Completed | 71 (Total number participants that are eligible and evaluable.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Total number eligible and evaluable
Arm/Group | Docetaxel Plus Trabectedin
Number analyzed (Participants) | 71
Age, Customized [Mean (Standard Deviation); unit: years] | 59.3 (9.2)
Age, Customized [Number; unit: participants]
  40-49 years | 10
  50-59 years | 28
  60-69 years | 25
  70-79 years | 7
  80-89 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 71
Cell Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 7
  Clear Cell Carcinoma | 3
  Endometrioid Adenocarcinoma | 6
  Mixed Epithelial Carcinoma | 2
  Serous Adenocarcinoma | 53

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumor Response
Description: Response is measured according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST v 1.0):
  Complete Response (CR) is disappearance of all target and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart.
  Partial Response (PR) is at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD.
  Disease Progression is at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD or the appearance of new lesions within 8 weeks of study entry.
  Stable Disease is any condition not meeting the above criteria.
  Indeterminate is defined as having no repeat tumor assessments following initiation of study therapy6
Time Frame: every other cycle for the first 6 months; then every 3 months thereafter (up to 5 years)
Population: Total number eligible and evaluable
Measure: Number; unit: participants
Arm/Group | Docetaxel Plus Trabectedin
Number analyzed (Participants) | 71
participants
  Partial response | 21
  Stable disease | 32
  Disease progression | 17
  Indeterminate | 1

2. Primary Outcome: Number of Participants With Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0
Time Frame: Prior to each cycle and 30 days after the last cycle (average of 5 months)
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel Plus Trabectedin
Number analyzed (Participants) | 71
Participants
  Leukopenia | 21
  Thrombocytopenia | 7
  Neutropenia | 21
  Anemia | 5
  Other hematologic | 2
  Constitutional | 8
  Nausea | 6
  Vomiting | 7
  Gastrointestinal | 11
  Hemorrhage | 1
  Infection | 10
  Metabolic | 10
  Musculoskeletal | 3
  Other neurological | 2
  Pain | 6
  Pulmonary | 2

3. Secondary Outcome: Duration of Progression-free Survival and Overall Survival
Time Frame: up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From study entry until disease progression or study withdrawal. Patients will then be monitored for delayed toxicity for a 5 year period.
Description: Activation through Mar 31, 2011, Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 (CTCAE v3.0) are utilized for defining and grading specific adverse events reported through the AdEERS system. Beginning Apr 1, 2011, CTCAE v 4.0 will be utilized for AE reporting through the AdEERS system. AEs are reported here using only CTCAEv3.0
Arm/Group | Docetaxel Plus Trabectedin
Serious Adverse Events (participants affected / at risk) | 31/71
Other Adverse Events (participants affected / at risk) | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Plus Trabectedin (N=71)
Tinnitus (Ear and labyrinth disorders) | 1
Neutrophils (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Obstruction, Gi - Ileum (Gastrointestinal disorders) | 2
Necrosis, Gi - Colon/Cecum/Appendix (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Gastrointestinal - Other (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hemorrhage, Gi - Rectum (Vascular disorders) | 1
Hemorrhage, Gi - Stomach (Vascular disorders) | 1
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1
Inf W/Gr 3 Or 4 Anc: Bladder (Urinary) (Infections and infestations) | 1
Edema: Head And Neck (Blood and lymphatic system disorders) | 1
Alt (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 2
Pain: Chest /Thorax Nos (General disorders) | 1
Pain: Back (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel Plus Trabectedin (N=71)
Rhinitis (Immune system disorders) | 2
Otitis Middle Ear (Ear and labyrinth disorders) | 1
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 5
Neutrophils (Blood and lymphatic system disorders) | 37
Platelets (Blood and lymphatic system disorders) | 43
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1
Leukocytes (Blood and lymphatic system disorders) | 40
Lymphopenia (Blood and lymphatic system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 70
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Ventricular Arrhythmia - Tachycardia (Cardiac disorders) | 1
S/N Arrhythmia: Sinus Tachycardia (Cardiac disorders) | 1
S/N Arrhythmia: Sinus Bradycardia (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 3
Hypotension (Cardiac disorders) | 4
Cardipulmonary Arrest (Cardiac disorders) | 1
International Normalized Ratio (Vascular disorders) | 1
Constitutional Symptoms - Other (General disorders) | 1
Sweating (General disorders) | 3
Weight Gain (General disorders) | 3
Fever (General disorders) | 10
Weight Loss (General disorders) | 8
Rigors/Chills (General disorders) | 6
Fatigue (General disorders) | 61
Insomnia (General disorders) | 10
Nail Changes (Skin and subcutaneous tissue disorders) | 6
Injection Site Reaction (Skin and subcutaneous tissue disorders) | 1
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 41
Induration (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Flushing (Skin and subcutaneous tissue disorders) | 5
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 6
Gastritis (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 9
Ascites (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 2
Distention (Gastrointestinal disorders) | 6
Taste Alteration (Gastrointestinal disorders) | 21
Incontinence, Anal (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 5
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 11
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 35
Anorexia (Gastrointestinal disorders) | 33
Dehydration (Gastrointestinal disorders) | 9
Constipation (Gastrointestinal disorders) | 32
Nausea (Gastrointestinal disorders) | 52
Diarrhea (Gastrointestinal disorders) | 40
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 2
Hemorrhage, Gi - Rectum (Vascular disorders) | 2
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 4
Hematoma (Vascular disorders) | 1
Hemorrhage, Gi - Abdomen Nos (Vascular disorders) | 1
Inf W/Gr 3 Or 4 Anc: Skin (Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Lung(Pneumonia) (Infections and infestations) | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Eye Nos (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Skin(Cellulitis) (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 8
Inf W/Nml Or Gr 1 Or 2 Anc: Abdomen Nos (Infections and infestations) | 1
Colitis, Infectious (Eg.C. Difficile) (Infections and infestations) | 2
Inf W/Gr 3 Or 4 Anc: Oral Cavity-Gums (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Vagina (Infections and infestations) | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Sinus (Infections and infestations) | 1
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 2
Inf W/Gr 3 Or 4 Anc: Pharynx (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 3
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 3
Edema: Limb (Blood and lymphatic system disorders) | 15
Edema: Head And Neck (Blood and lymphatic system disorders) | 1
Ast (Metabolism and nutrition disorders) | 18
Gfr (Metabolism and nutrition disorders) | 1
Metabolic/Laboratory - Other (Metabolism and nutrition disorders) | 6
Cholesterol,serum High (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 2
Hemoglobinuria (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Ggt (Metabolism and nutrition disorders) | 2
Alt (Metabolism and nutrition disorders) | 23
Alkaline Phosphatase (Metabolism and nutrition disorders) | 18
Bilirubin (Metabolism and nutrition disorders) | 3
Lipase (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 11
Hyperuricemia (Metabolism and nutrition disorders) | 2
Cpk (Metabolism and nutrition disorders) | 3
Bicarbonate, Serum-Low (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 19
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 22
Hypokalemia (Metabolism and nutrition disorders) | 18
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 16
Musculoskeletal/St: Other (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 9
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 7
Involuntary Movement (Nervous system disorders) | 3
Neurology - Other (Nervous system disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 10
Mood Alteration - Anxiety (Nervous system disorders) | 5
Mood Alteration - Agitation (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 1
Irritability (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 11
Neuropathy-Sensory (Nervous system disorders) | 33
Neuropathy-Motor (Nervous system disorders) | 2
Ocular/Visual - Other (Eye disorders) | 2
Dry Eye (Eye disorders) | 2
Flashing Lights/Floaters (Eye disorders) | 3
Blurred Vision (Eye disorders) | 11
Eyelid Dysfunction (Eye disorders) | 1
Pain - Other (General disorders) | 2
Pain: Urethra (General disorders) | 2
Pain: Chest /Thorax Nos (General disorders) | 4
Pain: Chest Wall (General disorders) | 5
Pain: Throat/Pharynx/Larynx (General disorders) | 3
Pain: Head/Headache (General disorders) | 16
Pain: Extremity-Limb (General disorders) | 3
Pain: Back (General disorders) | 11
Pain: Joint (General disorders) | 7
Pain: Bone (General disorders) | 7
Pain: Bladder (General disorders) | 2
Pain: Pain Nos (General disorders) | 2
Pain: Rectum (General disorders) | 3
Pain: Abdominal Pain Nos (General disorders) | 22
Pain: Cardiac/ Heart (General disorders) | 1
Pain: Tumor (General disorders) | 1
Pain: Liver (General disorders) | 1
Pain: Muscle (General disorders) | 7
Pulmonary: Other (Respiratory, thoracic and mediastinal disorders) | 2
Nasal/Paranasal Reactions (Respiratory, thoracic and mediastinal disorders) | 1
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27
Renal/Genitourinary - Other (Renal and urinary disorders) | 2
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Urinary Electrolyte Wasting (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 4
Renal Failure (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 5
Libido (Reproductive system and breast disorders) | 1
Vaginal Dryness (Reproductive system and breast disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No